CLINICAL TRIAL: NCT03477305
Title: BerryCare: A Blackberry Extension Lesson Series to Facilitate Community Engagement and Phytonutrient Intake
Brief Title: BerryCare: A Community Engagement Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dawn Brewer (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor-Investigator, Dawn Brewer, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 43452; P42ES007380 (NIH)
Record Dates: First submitted 2018-03-19; First posted 2018-03-26 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Cardiovascular Risk Factor
Keywords: older adults; community gardening; cooperative extension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BerryCare Participants (Experimental): Subjects will be recruited to participate in a community gardening program where they will learn the benefits of both physical active gardening and consuming homegrown foods through blackberry consumption.
  Interventions: Behavioral: Blackberry Consumption

INTERVENTIONS:
Behavioral: Blackberry Consumption — Measures of biomedical and behavioral changes resulting from the consumption of blackberries.

SUMMARY:
BerryCare teaches people about the health benefits of blackberries, how to harvest and maintain blackberry bushes and then assesses changes in knowledge and behaviors associated with blackberries and physical measurements.

DETAILED DESCRIPTION:
BerryCare seeks to teach community members how to grow thornless, erect blackberry brambles and to healthily consume fresh blackberries using Plate It Up Kentucky Proud recipes. Horticulture, nutrition, and extension experts are working together to design a blackberry-growing program that engages citizens and their community in each step of the process, from planting to harvesting berries. The lessons will be delivered by experts in their respective field, with accompanying extension publications and supplemental materials provided for replication of the curriculum in other counties.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older

Exclusion Criteria:

* Physically incapacitated
* Mentally incapacitated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-01-18 (Actual); Primary Completion 2018-09-26 (Actual); Study Completion 2018-09-26 (Actual)

PRIMARY OUTCOMES:
Change in consumption of blackberries | Baseline, 6 months, 12 months, 18 months
  Blackberry consumption will be measured in participants during pre screening and throughout the course of the study.

SECONDARY OUTCOMES:
Change in blood pressure | Baseline, 6 months, 12 months, 18 months
  The effect of blackberry consumption on blood pressure will be assessed at baseline and throughout the study.
Change in total cholesterol | Baseline, 6 months, 12 months, 18 months
  The effect of blackberry consumption on total cholesterol will be assessed at baseline and throughout the study.
Change in HDL cholesterol | Baseline, 6 months, 12 months, 18 months
  The effect of blackberry consumption on HDL cholesterol will be assessed at baseline and throughout the study.
Change in LDL cholesterol | Baseline, 6 months, 12 months, 18 months
  The effect of blackberry consumption on LDL cholesterol will be assessed at baseline and throughout the study.
Change in A1c | Baseline, 6 months, 12 months, 18 months
  The effect of blackberry consumption on A1c will be assessed at baseline and throughout the study.
Change in carotenoids | Baseline, 6 months, 12 months, 18 months
  The effect of blackberry consumption on carotenoid status will be assessed at baseline and throughout the study.
Change in weight | Baseline, 6 months, 12 months, 18 months
  The effect of blackberry consumption on weight will be assessed at baseline and throughout the study.
Change in waist circumference | Baseline, 6 months, 12 months, 18 months
  The effect of blackberry consumption on waist circumference will be assessed at baseline and throughout the study.
Change in knowledge | Baseline, 6 months, 12 months, 18 months
  The effect of blackberry consumption on knowledge of phytonutrients and recommended servings of fruits and vegetables will be assessed at baseline and throughout the study.
Change in self-reported fruit and vegetable intake | Baseline, 6 months, 12 months, 18 months
  The effect of blackberry consumption on self-reported fruit and vegetable intake will be assessed at baseline and throughout the study.
Change in group cohesion | Baseline, 6 months, 12 months, 18 months
  The effect of blackberry consumption on group cohesion will be assessed at baseline and throughout the study.
Change in physical function | Baseline, 6 months, 12 months, 18 months
  The effect of blackberry consumption on physical function will be assessed at baseline and throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Brewer, PhD, Principal Investigator — University of Kentucky
Locations (5):
- United States (5):
  - Red Bird Mission, Beverly, Kentucky
  - Harlan County Extension Office, Harlan, Kentucky
  - University of Kentucky, Lexington, Kentucky
  - Jessamine County Senior Citizens Center, Nicholasville, Kentucky
  - Cowan Community Center, Whitesburg, Kentucky

IPD SHARING:
Plan to Share IPD: No
No plan to share data.